CLINICAL TRIAL: NCT07024043
Title: Effect of Dexamethasone Versus Dexmedetomidine as A Local Anesthetic Adjuvant In IPACK Block for Post Operative Analgesia Following Arthroscopic Knee Surgeries
Brief Title: Dexamethasone Versus Dexmedetomidine in IPACK Block to Reduce Pain Post Arthroscopic Knee Surgeries
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU MS 173/2025
Record Dates: First submitted 2025-05-06; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-03

CONDITIONS: Efficacy of Drugs in Pain Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- (Group 1) for iPACK block with 0.25% bupivacaine only. (Group 2) for iPACK block with 0.25% bupivac (Experimental): For each group, patients will be put in supine position, the procedure will be performed under complete aseptic precautions and All patients will be divided into three groups:(Group 1) for iPACK block with 0.25% bupivacaine only. (Group 2) for iPACK block with 0.25% bupivacaine and dexamthasone and (Group 3) for iPACK block with 0.25% bupivacaine and dexmedetomidine .
  Interventions: Drug: Dexamethasone versus Dexmedetomidine in IPACK Block to reduce pain post Arthroscopic knee surgeries; Procedure: IPACK and multi-modal analgesic regimen

INTERVENTIONS:
Drug: Dexamethasone versus Dexmedetomidine in IPACK Block to reduce pain post Arthroscopic knee surgeries — Blocks will be carried out with the patient supine with the operative leg externally rotated and slightly flexed at the knee or in prone position.with Ultrasound device with a high-frequency (6-13 MHz) linear probe using in plane lateral to medial approach and this will be done by a senior staff anaesthesia physician skilled in ultrasound guided regional anaesthesia.
Procedure: IPACK and multi-modal analgesic regimen — patients will be put in supine position, the procedure will be performed under complete aseptic precautions and All patients will be divided into three groups:(Group 1) for iPACK block with 0.25% bupivacaine only. (Group 2) for iPACK block with 0.25% bupivacaine and dexamthasone and (Group 3) for iPACK block with 0.25% bupivacaine and dexmedetomidine .

SUMMARY:
The investigators will test the effects of dexamethasone versus dexmedetomidine as adjuvant to bupivacaine in IPACK Block and it's direct effect in decreasing pain post operative following Arthroscopic knee surgeries

DETAILED DESCRIPTION:
A.Preoperative settings: All patients will be assessed preoperatively by careful history taking, full physical examination, and laboratory evaluation. An informed written consent will be taken from every patient just before the surgery. B.Intraoperative and postoperative settings: On arrival to the operating room, baseline parameters such as ECG, mean arterial blood pressure, heart rate, and oxygen saturation will be recorded. Intravenous line will be inserted and IV Ringer's solution will be started, 500ml bolus will be given as a preload over 20 min before performing spinal anaesthesia and maintenance volume of 10ml\kg. For each group, patients will be put in supine position, the procedure will be performed under complete aseptic precautions and All patients will be divided into three groups:(Group 1) for iPACK block with 0.25% bupivacaine only. (Group 2) for iPACK block with 0.25% bupivacaine and dexamthasone and (Group 3) for iPACK block with 0.25% bupivacaine and dexmedetomidine .

ELIGIBILITY:
Inclusion Criteria:

* Physical status: ASA I,II. Both sexes. BMI<35

Exclusion Criteria:

* Refusal of the procedure or participation in the study by the patient. Physical status: ASA III or Above. History of allergy to the study drug. Evidence of local infection at site of injection. Major hepatic, renal, or cardiovascular dysfunction. BMI>35.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Dexamethasone versus Dexmedetomidine in IPACK Block to reduce pain post Arthroscopic knee surgeries | 45 minutes after spinal anaesthesia
  postoperative analgesic effect will be assessed by the time till first analgesic requirement which is defined as the time (in hours) after finishing of ultrasound guided iPACK block till the patient's requirement for first analgesia postoperative in ward.
  Postoperative pain will be assessed by visual analog scale (VAS) up to 24 h after surgery. Whenever VAS score reached ≥ 4, rescue analgesia will be given in the form of iv injection diclofenac sodium 75 mg. Time to the first dose of diclofenac sodium postoperatively will be recorded

SECONDARY OUTCOMES:
Effect Of Dexamethasone Versus Dexmedetomidine as A Local Anesthetic Adjuvant In IPACK Block for Post Operative Analgesia following Arthroscopic Knee Surgeries | 45 minutes after spinal anesthesia
  Total analgesics consumption (in mg.) over 24-hour period post-operative.
  Incidence of adverse effects such as:
  Hematoma, hypotension (considered as significant hypotension when blood pressure decrease by 20% relative to baseline), bradycardia (considered as significant bradycardia when heart rate decrease by 20% relative to baseline), nausea and/or vomiting, local anesthetic toxicity, post operative paresthesia, sedation (assessed by Ramsay sedation score) and hypoxemia (Spao2<90%) will be recorded in both groups and will be properly managed by fluid reuscitation, oxygen support, vasopressor and proton pump inhibitors.
  Post-operative ambulation enhancement in the form of: time of start of ambulation (in hours) starting from end of surgery- walking- climbing stairs (according to the New Knee Society Knee Scoring System)

CONTACTS AND LOCATIONS:
Overall Officials: Maisa Essam Abdelhaleem, MBBCH, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Time Frame: Before 1/2026
Access Criteria: Free